CLINICAL TRIAL: NCT04409275
Title: STUDY OF THE APPEARANCE OF LUNG FIBROTIC CHANGES ASSOCIATED WITH SARS-CoV-2 INFECTION
Brief Title: LUNG FIBROTIC CHANGES ASSOCIATED WITH SARS-CoV-2 INFECTION
Acronym: INC-CVD-202001
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: INC-CVD-2020-01
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, observational, multicenter study that will evaluate the changes in lung function that patients admitted with SARS-CoV-2 pneumonia will present according to the level of severity at 4, 12, 26 and 52 weeks after hospital discharge.

DETAILED DESCRIPTION:
The project consists of a prospective, observational, multicenter study that will evaluate changes in lung function (forced spirometry, measurement of static lung volumes using plethysmography and pulmonary carbon monoxide diffusion test) that patients admitted with pneumonia will present. caused by SARS-CoV-2 according to the level of severity at 4, 12, 26 and 52 weeks after discharge from hospital. Restrictive pulmonary abnormalities will be confirmed by imaging tests (high resolution chest CT).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for bilateral pneumonia caused by SARS-CoV-2 (confirmed by PCR).
* Age over 18 years.
* Acceptance of informed consent.
* Life expectancy over 1 year.

Exclusion Criteria:

* Patients with a previous diagnosis of interstitial lung disease.
* Inability to attend review visits.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with pneumonia caused by SARS-CoV-2
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary fibrotic changes, short and medium term | 12 months
  To analyze the number of patients who will develop pulmonary fibrotic changes, in the short and medium term, after surviving a bilateral pulmonary infection by SARS-CoV-2
Degree of lung function impairment | 6 and 12 months
  To study the degree of lung function impairment, specifically the restrictive changes in functional capacity and diffusion alterations and its relationship with clinical variables.
Biological markers | 1 month
  Examine the biological markers in the patients who will present this dysregulation of the curative response that will give rise to pulmonary fibrosing phenomena.

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Department. Hospital Clinico., Valencia, Spain

REFERENCES:
- [Derived] Gonzalez-Villaescusa C, Tarraso Castillo J, Martinez-Pitarch D, Riesco Miranda JA, Garcia-Castillo E, Gotera Rivera C, Carrasco Hernandez L, Sobradillo Ecenarro P, Signes-Costa J, Naval Sendra E, Callejas Gonzalez FJ, Yordi Leon A, Vigil Gimenez L, Nunez Fernandez M, Palop Cervera M, Carbonell-Asins JA, Agusti A; Field Investigators. Predictors of Progression in Pre-COPD: The 3P Study Rationale and Design. Open Respir Arch. 2025 Nov 17;8(1):100519. doi: 10.1016/j.opresp.2025.100519. eCollection 2026 Jan-Mar. PMID 41438363
- [Derived] Botello-Marabotto M, Tarraso J, Mulet A, Presa-Fernandez L, Fernandez-Fabrellas E, Portal JAR, Ros JA, Lozano-Vicente D, Bernardos A, Martinez-Bisbal MC, Martinez-Manez R, Signes-Costa J. Metabolomic Biomarkers of Pulmonary Fibrosis in COVID-19 Patients One Year After Hospital Discharge. J Med Virol. 2025 Mar;97(3):e70289. doi: 10.1002/jmv.70289. PMID 40088077
- [Derived] Tarraso J, Safont B, Carbonell-Asins JA, Fernandez-Fabrellas E, Sancho-Chust JN, Naval E, Amat B, Herrera S, Ros JA, Soler-Cataluna JJ, Rodriguez-Portal JA, Andreu AL, Marin M, Rodriguez-Hermosa JL, Gonzalez-Villaescusa C, Soriano JB, Signes-Costa J; COVID-FIBROTIC study team. Lung function and radiological findings 1 year after COVID-19: a prospective follow-up. Respir Res. 2022 Sep 12;23(1):242. doi: 10.1186/s12931-022-02166-8. PMID 36096801
- [Derived] Safont B, Tarraso J, Rodriguez-Borja E, Fernandez-Fabrellas E, Sancho-Chust JN, Molina V, Lopez-Ramirez C, Lope-Martinez A, Cabanes L, Andreu AL, Herrera S, Lahosa C, Ros JA, Rodriguez-Hermosa JL, Soriano JB, Moret-Tatay I, Carbonell-Asins JA, Mulet A, Signes-Costa J. Lung Function, Radiological Findings and Biomarkers of Fibrogenesis in a Cohort of COVID-19 Patients Six Months After Hospital Discharge. Arch Bronconeumol. 2022 Feb;58(2):142-149. doi: 10.1016/j.arbres.2021.08.014. Epub 2021 Sep 3. PMID 34497426